CLINICAL TRIAL: NCT02703480
Title: Comparison of d-PTFE Membrane With Titanium-mesh in Vertical Ridge Augmentation: A Split Mouth, Randomized Controlled Clinical Trial
Brief Title: Comparing the Efficacy and Morbidity of Two Vertical Ridge Augmentation Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11877
Record Dates: First submitted 2015-11-06; First posted 2016-03-09 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Vertical Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- All Study Participants - d-PTFE (Experimental): The proposed study design is a randomized controlled trial, split mouth design, to compare the two different vertical augmentation procedures: Titanium mesh (Ti-mesh) technique and Guided Bone Regeneration (GBR) technique with a high-density polytetrafluoroethylene (d-PTFE) membrane.
  Interventions: Biological: d-PTFE
- All Study Participants - Ti-mesh (Experimental): The proposed study design is a randomized controlled trial, split mouth design, to compare the two different vertical augmentation procedures: Titanium mesh (Ti-mesh) technique and Guided Bone Regeneration (GBR) technique with a high-density polytetrafluoroethylene (d-PTFE) membrane
  Interventions: Biological: Ti-mesh

INTERVENTIONS:
Biological: d-PTFE — high-density polytetrafluoroethylene (d-PTFE) membrane
  Arms: All Study Participants - d-PTFE
Biological: Ti-mesh — Titanium mesh
  Arms: All Study Participants - Ti-mesh

SUMMARY:
The proposed study design is a randomized controlled trial, split mouth design, to compare the two different vertical augmentation procedures: Titanium mesh (Ti-mesh) technique and Guided Bone Regeneration (GBR) technique with a high-density polytetrafluoroethylene (d-PTFE) membrane.

DETAILED DESCRIPTION:
E) Study Procedures Visit 1: Screening (Approximately 30 mins) Informed consent will be obtained by the principal investigator or a co-investigator. The subjects will be instructed to read the informed consent form (ICF), given ample time to have any questions answered, and then instructed to sign the ICF. Subject will be given a copy of the ICF.

Subject will be asked to complete demographic information and a medical history.

Inclusion/exclusion criteria will be evaluated.

The pre-operative height of the bony crest will be evaluated on the pre-existing radiographs from the referring clinic if they are less than 6 months old. If recent radiographs do not exist, radiographs will be taken at this visit. It is standard of care to have radiographs from within the past 6 months prior to surgery.

Visit 2: Surgery (Approximately 180 mins) Medical history will be reviewed as standard of care. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.

Surgeries will be performed by either of two investigators, Yong Hur (Co-I) and Yumi Ogata (PI).

The use of d-PTFE for vertical ridge augmentation will be randomly assigned to one side of the mouth of each subject (randomization is for research purposes) and Ti-mesh to the other side of mouth, and therefore, subjects will receive both of the following procedures:

* Guided Bone regeneration (GBR) procedure using a d-PTFE: (standard of care excluding clinical measurements) The following steps will be performed following standard of care procedures: local anesthesia, muco-periosteal incision, full thickness flap reflection, de-cortication of the alveolar ridge, bone harvesting using bone scrapers, tenting screw placement, clinical measurements, DBBM graft material placement, the placement and stabilization of the d-PTFE membrane according to manufacturer's instructions, sutures.
* Guided Bone regeneration (GBR) procedure using Ti-mesh: (standard of care excluding clinical measurements) The following steps will be performed following standard of care procedures: local anesthesia, muco-periosteal incision, full thickness flap reflection, de-cortication of the alveolar ridge, bone harvesting using bone scrapers, tenting screw placement, clinical measurements, DBBM graft material placement, the placement and stabilization of the titanium mesh according to manufacturer's instructions, sutures.

Bone harvesting using bone scrapers will be performed during GBR procedures with both techniques (d-PTFE and Ti-mesh). Bone harvesting using bone scrapers is for harvesting particulate autogeneous bone graft material. The investigators will use a mixture of 50:50 DBBM and autogenous bone graft material for all vertical augmentation procedures in the study. Particulate autogenous bone graft will be harvested from the retromolar region of the mandible. This area is just next to the area of GBR procedures (posterior mandible) and will be visible after flap elevation for vertical augmentation. Therefore, the investigators do not need any additional steps except harvesting autogenous bone graft. Intraoral harvesting by bone scrapers from the retromolar region is a simple and safe method for collecting cortical bone chips.

The intrasurgical clinical measurements of the ridge height will be taken during surgery. The distance between the top of the tenting screw and bone crest will be measured with a periodontal probe during the procedure. Duration of each procedure and surgical complications including flap tear and bleeding will be collected. All outcome measurements will be performed by a Co-I who did not perform the surgery.

The subject will be asked to complete a pain/discomfort survey using VAS scale from zero to ten. A medication log will be given to the patient to track the number of pills of the prescribed painkiller they have taken in order to examine the amount of pain after the surgical procedures. The mean number of pills used after surgical procedures will be analyzed.

Post-operative medication will be prescribed following TUSDM standard of care guidelines.

Visit 3 (7±3 days after procedure): Post-operative Follow-up (Approximately 20 mins)

Medical history will be reviewed as standard of care. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.

Each subject will have a post-operative visit, which is standard practice at TUSDM periodontology clinic. Standard of care procedures including suture removal and evaluation of surgical site will be performed.

For research, information regarding bleeding, presence of infection, bruising, and/or other complications will be collected. Each subject will complete a survey to evaluate the level of pain/discomfort, bleeding, and swelling following the surgical procedure for each side - each classified on a VAS scale from zero to ten. In addition, the subject will return his or her completed medication log.

Visit 4 (21±3 days after procedure): Post-operative Follow-up (Approximately 20 mins)

Medical history will be reviewed as standard of care. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.

Each subject will have a post-operative visit, which is standard practice at TUSDM periodontology clinic. Standard of care procedures including suture removal and evaluation of surgical site will be performed.

For research, information regarding bleeding, presence of infection, bruising, and/or other complications will be collected. Each subject will complete a survey to evaluate the level of pain/discomfort, bleeding, and swelling following the surgical procedure for each side - each classified on a VAS scale from zero to ten.

Follow-up visits during the six month post-operative period of the vertical ridge augmentation surgery will be scheduled. Standard of care procedures and evaluations will be completed during follow-up visits. The surgical sites will be evaluated after the vertical ridge augmentation procedures, in order to assess the presence of postoperative complications, such as the exposure of a d-PTFE membrane or Ti-mesh, infection, swelling, paresthesia or any other complications. All will be noted in the subject's axiUm record and reviewed at the time of Visit 4.

Visit 5 (6±1 months after Visit 4): Evaluation visit (Approximately 20 mins) Medical history will be reviewed as standard of care. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.

Surgical sites will be evaluated and the subject's axiUm record will be reviewed for any complications.

Each subject will complete a survey to evaluate the level of pain/discomfort, bleeding, and swelling following the surgical procedure for each side - each classified on a VAS scale from zero to ten, as at Visit 3.

Radiographs will be taken. It is standard of care to have radiographs taken prior to implant placement. The post-operative (after the vertical GBR augmentation procedure) height of the bony crest will be evaluated on the radiographs taken as part of standard of care.

Visit 6 (Up to 1 month after Visit 5): Bone core harvesting, implant placement visit (Approximately 120 mins) Medical history will be reviewed as standard of care. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.

The subject will present for their regularly scheduled implant placement. The following steps will be performed following standard of care procedures: local anesthesia, muco-periosteal incision, full thickness flap reflection, membrane (Ti-mesh/d-PTFE) removal, clinical measurements, tenting screws removal, bone core harvesting, implant osteotomy, implant placement, and sutures.

The intrasurgical clinical measurements of the ridge height will be taken at during implant placement surgery. The distance between the top of the tenting screw and bone crest will be measured with a periodontal probe during the procedure. The bone height gain will be calculated by subtracting the second measurement form the first measurement (taken during initial surgery).

At the time of the implant placement a bone core will be harvested from each site of the implant locations for histological analysis. For the bone samples in this study, a hollow (trephine) bur, rather than solid bur, will be used to allow for sampling. A trephine bur with 3-4 mm diameter will be used. The core size will not exceed the amount of bone removal required for designated implants. Removal of bone is standard during implant placement in order to create space for the fixture.

The bone core biopsies will be placed in fixative and labeled with subject ID. The collected bone samples will be placed in alcohol for storage and stored in a basic science laboratory DHS-635.

The implant placement will not be considered a part of this study.

After Visit 6 - Laboratory analysis of bone core sample Histological slides will be prepared and histomorphometric analysis will be performed by the commercial laboratory (CBSET). The samples will be coded as subject numbers and histological analysis will be blinded. All collected bone core samples will be shipped to the laboratory (CBSET) by Yumi Ogata (PI) or Yong Hur (Co-I).

Histomorphometric measurements of the tissue fractions (DBBM, autogenous bone, newly formed bone and marrow and/or connective tissue) will be performed for the grafted area. The sections will be digitally photographed with computerized software.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Non-smokers
* Existence of bilateral vertical/horizontal ridge deformities (Seibert Class III)
* The length of the edentulous span is from two or more teeth

Exclusion Criteria:

* The patients will not be admitted in the study if any of the following exclusion criteria are met:

  * Patients who have an infectious disease (self reported - HIV, tuberculosis or hepatitis)
  * Known allergies to the research-related materials
  * Patients who have compromised healing potential:
* bone metabolic disease e.g., Paget's disease, osteoporosis, osteomalacia
* uncontrolled diabetes: HbA1c >=7, values measured within six months (using the existing record in AxiUm or if the subject has the condition, but there is no report in AxiUm - a blood test record will be requested)
* patient currently taking steroid medication
* history of oral bisphosphonate intake greater than 3 years or any IV administration

  * Pregnant or lactating patients (self-reported), as part of TUSDM standard of care not to treat for non-emergency surgical procedures
  * Presence of surgical scar tissue from previous surgical procedure in the posterior mandible
  * Pathology present within the alveolar ridges in the posterior mandible, determined clinically or radiographically
  * History of radiation therapy to the mandible
  * Smokers
* Elective periodontal procedures are postponed during pregnancy, active infectious disease, bisphosphonate intake or uncontrolled diabetes as standard of care in the TUSDM department of periodontology. Diseases or conditions which have been shown to affect healing are excluded for research. Vertical ridge augmentation is not contraindicated with pregnancy and there is no known safely issues associated with it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2025-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yumi Ogata, DMD, DDS, MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 participants were enrolled for a split-mouth study. 10 participants completed the study (20 sites).
Units Other Than Participants: Sites
Period: Overall Study
Arm/Group | All Study Participants - d-PTFE | All Study Participants - Ti-mesh
Started | 11; 11 Sites | 11; 11 Sites
Completed | 10; 10 Sites | 10; 10 Sites
Not Completed | 1; 1 Sites | 1; 1 Sites

BASELINE CHARACTERISTICS:
Population: A total of 11 participants were enrolled for a split-mouth study. Each participant had two research sites and each of two treatments are randomly assigned to either the right or left side of mandible. A total of 10 patients (20 sites) completed all study visits and were included in analysis.
Groups:
- All Study Participants: The proposed study design is a randomized controlled trial, split mouth design, to compare the two different vertical augmentation procedures: Titanium mesh (Ti-mesh) technique and Guided Bone Regeneration (GBR) technique with a high-density polytetrafluoroethylene (d-PTFE) membrane
  Ti-mesh: Titanium mesh
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.058)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Vertical defect height (mm) at measured at baseline [Mean (Standard Deviation); unit: millimeter] | 4.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Vertical Bone Height
Description: intrasurgical clinical measurement in millimeter
Time Frame: from 6 months to 8 months following the procedure
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | All Study Participants - d-PTFE | All Study Participants - Ti-mesh
Number analyzed (Participants) | 10 | 10
millimeter | 3.7 (1.2) | 3.2 (1.1)

2. Secondary Outcome: Rate of Post-Operative Complications
Description: compare the rate of post-operative complications over the six months healing period after vertical augmentation procedures
Time Frame: Up to 6 months to 8 months following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants - d-PTFE | All Study Participants - Ti-mesh
Number analyzed (Participants) | 10 | 10
Participants | 2 | 2

3. Secondary Outcome: Bone Core Histology
Description: Histomorphometric measurements of the tissue fractions (newly formed bone, DBBM, autogenous bone, and marrow and/or connective tissue) will be performed for the grafted area.
Time Frame: from 6 months to 8 months following the procedure
Reporting Status: Not Posted, anticipated posting 2025-03

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | All Study Participants - d-PTFE | All Study Participants - Ti-mesh
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants - d-PTFE (N=10) | All Study Participants - Ti-mesh (N=10)
Membrane exposure (Injury, poisoning and procedural complications) | 1 | 2
abscess (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02703480/Prot_SAP_000.pdf